CLINICAL TRIAL: NCT00945009
Title: Treatment for Patients With Bilateral, Multicentric, or Bilaterally-Predisposed Unilateral Wilms Tumor
Brief Title: Combination Chemotherapy and Surgery in Treating Young Patients With Wilms Tumor
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AREN0534; NCI-2011-01953 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000649716; AREN0534 (Other: Children's Oncology Group); AREN0534 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Adult Kidney Wilms Tumor; Beckwith-Wiedemann Syndrome; Childhood Kidney Wilms Tumor; Diffuse Hyperplastic Perilobar Nephroblastomatosis; Rhabdoid Tumor of the Kidney; Stage I Kidney Wilms Tumor; Stage II Kidney Wilms Tumor; Stage III Kidney Wilms Tumor; Stage IV Kidney Wilms Tumor; Stage V Kidney Wilms Tumor
MeSH Terms: conditions — Wilms Tumor; Beckwith-Wiedemann Syndrome | interventions — Dactinomycin; Doxorubicin; Radiotherapy; Radiation; Vincristine

ARMS (3):
- Arm 1 (Bilateral Wilms Tumors) (Experimental): Patients start with three drug chemotherapy (Regimen VAD; vincristine, dactinomycin and doxorubicin) and are evaluated and six and 12 weeks for feasibility of undergoing a partial nephrectomy/renal sparing surgery. At week 12 definitive surgery takes place followed by chemotherapy and radiation therapy based on histology and stage. Treatment continues for 25 or 31 weeks depending on histology. Patients are followed for up to 10 years following end of therapy.
  Interventions: Biological: Dactinomycin; Drug: Doxorubicin Hydrochloride; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery; Drug: Vincristine Sulfate
- Arm 2 (Unilateral High Risk tumors bilaterally predisposed) (Experimental): Patients start with either 2 drug or three drug chemotherapy (Regimen VA, VAD) and are evaluated a 6 and 12 weeks for feasibility of undergoing a partial nephrectomy. At week 12 definitive surgery takes place followed by chemotherapy.
  Interventions: Biological: Dactinomycin; Drug: Doxorubicin Hydrochloride; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery; Drug: Vincristine Sulfate
- Arm 3 (DHPLN) (Experimental): Patients with this rare disease are diagnosed based on cross-sectional imaging characteristics and undergo 2 drug chemotherapy (Regimen;VA). Patients are reassessed at 6 weeks and 12 weeks. If disease has responded or stayed stable chemotherapy is completed for 19 weeks (Regimen EE4A). If disease has progress a biopsy is performed to assess histology and adjust therapy based on the biopsy. This therapy may include, nephrectomy, chemotherapy or radiation therapy.
  Interventions: Biological: Dactinomycin; Drug: Doxorubicin Hydrochloride; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery; Drug: Vincristine Sulfate

INTERVENTIONS:
Biological: Dactinomycin — Given IV
  Other Names: Actinomycin A IV; Actinomycin C1; Actinomycin D; Actinomycin I1; Actinomycin IV; Actinomycin X 1; Actinomycin-[thr-val-pro-sar-meval]; Cosmegen; DACT; Dactinomycine; Lyovac Cosmegen; Meractinomycin
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase III trial studies how well combination chemotherapy and surgery work in treating young patients with Wilms tumor. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving it after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To improve 4-year event-free survival (EFS) to 73% for young patients with bilateral Wilms tumor (BWT).

II. To prevent complete removal of at least one kidney in 50% of patients with BWT by using prenephrectomy 3-drug chemotherapy induction with vincristine (vincristine sulfate), dactinomycin, and doxorubicin (doxorubicin hydrochloride).

III. To evaluate the efficacy of chemotherapy in preserving renal units in children with diffuse hyperplastic perilobar nephroblastomatosis (DHPLN) and preventing Wilms tumor development.

IV. To facilitate partial nephrectomy in lieu of nephrectomy in 25% of children with unilateral tumors and aniridia, Beckwith-Wiedemann syndrome (BWS), hemihypertrophy or other overgrowth syndromes, by using prenephrectomy 2-drug chemotherapy induction with vincristine and dactinomycin.

V. To have 75% of patients with BWT undergo definitive surgical treatment by 12 weeks after initiation of chemotherapy.

OUTLINE: Patients are assigned to 1 of 3 arms.

ARM 1 (Bilateral Wilms Tumors): Patients start with three drug chemotherapy (Regimen VAD; vincristine, dactinomycin and doxorubicin) and are evaluated and six and 12 weeks for feasibility of undergoing a partial nephrectomy/renal sparing surgery. At week 12 definitive surgery takes place followed by chemotherapy and radiation therapy based on histology and stage. Treatment continues for 25 or 31 weeks depending on histology. Patients are followed for up to 10 years following end of therapy.

ARM 2 (Unilateral High Risk tumors bilaterally predisposed): Patients start with either 2 drug or three drug chemotherapy (Regimen VA, VAD) and are evaluated a 6 and 12 weeks for feasibility of undergoing a partial nephrectomy. At week 12 definitive surgery takes place followed by chemotherapy.

ARM 3 (DHPLN): Patients with this rare disease are diagnosed based on cross-sectional imaging characteristics and undergo 2 drug chemotherapy (Regimen;VA). Patients are reassessed at 6 weeks and 12 weeks. If disease has responded or stayed stable chemotherapy is completed for 19 weeks (Regimen EE4A). If disease has progress a biopsy is performed to assess histology and adjust therapy based on the biopsy. This therapy may include, nephrectomy, chemotherapy or radiation therapy.

VAD REGIMEN: Patients receive vincristine sulfate intravenously (IV) over 1 minute on days 1, 8, 15, 22, 29, and 36 (weeks 1-6) and dactinomycin IV and doxorubicin hydrochloride IV over 15-120 minutes on days 1 and 22 (weeks 1 and 4).

EE4A REGIMEN: Patients receive vincristine sulfate IV over 1 minute on days 1, 8, 15, 22, 29, and 36 (weeks 1-6) and dactinomycin IV over 1-5 minutes on days 1 and 22 (weeks 1 and 4).

After completion of study treatment, patients are followed up periodically for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have one of the following conditions to be eligible:

  * Synchronous bilateral Wilms tumors**; or
  * Unilateral Wilms tumor and aniridia, Beckwith-Wiedemann Syndrome, idiopathic hemihypertrophy, Simpson-Golabi-Behmel-Syndrome, Denys-Drash Syndrome or other associated genitourinary anomalies associated with bilateral Wilms tumor, such as hypospadias and undescended testis (to be eligible, these patients must not undergo any nephrectomy at diagnosis; note-horseshoe kidney is not associated with bilateral Wilms tumor and these patients should go on the appropriate unilateral Wilms tumor study); or
  * Multicentric Wilms tumor (any age) (to be eligible, these patients must not undergo any nephrectomy at diagnosis); or
  * Unilateral Wilms tumor with contralateral nephrogenic rest(s) (any size) in a child under one year of age (to be eligible, these patients must not undergo any nephrectomy at diagnosis); or
  * Diffuse hyperplastic perilobar nephroblastomatosis (unilateral or bilateral) defined by central radiological review; or
  * Wilms tumor arising in a solitary kidney (patients with metachronous Wilms tumor are not eligible)

    * The AREN0534 study uses the guideline that Wilms tumor with a single lesion 1 cm or greater in the contralateral kidney or multiple lesions (of any size) in the contralateral kidney should be treated on the synchronous bilateral Wilms tumor stratum; patients with an isolated lesion less than 1 cm in the contralateral kidney should be treated on the appropriate study for unilateral Wilms tumor OR on the unilateral Wilms tumor/contralateral nephrogenic rest stratum of this study if they have not undergone nephrectomy and are under one year of age
  * Loss of heterozygosity (LOH) results-which are used in the unilateral Wilms tumor studies-are not a requirement for enrollment on AREN0534; blood samples can be submitted but will not be used to direct AREN0534 therapy
* Specimens/materials must be submitted for central review by day 7; for enrollment on AREN0534, unless a biopsy was done, the submission requirements at enrollment on AREN03B2 refer to imaging studies; tissue samples are only required if a surgical procedure (biopsy or nephrectomy) was performed at the time of enrollment on AREN03B2
* Patients must begin protocol therapy on AREN0534 by day 14 following surgery or diagnosis by initial computed tomography (CT)/magnetic resonance imaging (MRI), unless medically contraindicated
* Karnofsky performance status must be >= 50% for patients > 16 years of age and Lansky performance status must be >= 50% (for patients =< 16 years of age
* Patients must not have received systemic chemotherapy or radiation therapy prior to treatment on this study
* Patients with unilateral Wilms tumor and aniridia, Beckwith-Wiedemann Syndrome, idiopathic hemihypertrophy, Simpson-Golabi-Behmel-Syndrome, Denys-Drash Syndrome or other associated genitourinary anomalies; or multicentric or unilateral Wilms tumor with contralateral nephrogenic rest(s) (any size) in a child under 1 year of age who undergo a nephrectomy at diagnosis are not eligible for this study and should be directed to a unilateral Wilms tumor study
* Total bilirubin =< 1.5 times upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 times upper limit of normal (ULN) for age
* Shortening fraction >= 27% by echocardiogram, OR ejection fraction >= 50% by radionuclide angiogram

  * (Cardiac function does not need to be assessed in patients who will not receive doxorubicin as part of their initial therapy on this study [i.e., patients who start on regimen EE-4A])
* Female patients of childbearing age must have a negative pregnancy test
* Female patients who are lactating must agree to stop breastfeeding
* Sexually active patients of childbearing potential must agree to use effective contraception
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met
* No concurrent aprepitant

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 249 (Actual)
Dates: Start 2009-07-13 (Actual); Primary Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter F Ehrlich, Principal Investigator — Children's Oncology Group
Locations (169):
- United States (146):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Schneider Children's Medical Center of Israel, Petah Tikua, Israel
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Ehrlich PF, Tornwall B, Chintagumpala MM, Chi YY, Hoffer FA, Perlman EJ, Kalapurakal JA, Warwick A, Shamberger RC, Khanna G, Hamilton TE, Gow KW, Paulino AC, Gratias EJ, Mullen EA, Geller JI, Fernandez CV, Dome JS. Kidney Preservation and Wilms Tumor Development in Children with Diffuse Hyperplastic Perilobar Nephroblastomatosis: A Report from the Children's Oncology Group Study AREN0534. Ann Surg Oncol. 2022 May;29(5):3252-3261. doi: 10.1245/s10434-021-11266-6. Epub 2022 Jan 24. PMID 35072864
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 (Bilateral Wilms Tumors) | Arm 2 (Unilateral High Risk Tumors Bilaterally Predisposed) | Arm 3 (DHPLN)
Started | 201 | 39 | 9
Completed | 156 | 32 | 6
Not Completed | 45 | 7 | 3
Not completed — Lack of Efficacy | 10 | 0 | 0
Not completed — Physician Decision | 21 | 4 | 3
Not completed — Protocol Violation | 6 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Ineligible | 6 | 1 | 0
Not completed — Inevaluable | 0 | 1 | 0
Not completed — Refusal of further protocol | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Bilateral Wilms Tumors) | Arm 2 (Unilateral High Risk Tumors Bilaterally Predisposed) | Arm 3 (DHPLN) | Total
Number analyzed (Participants) | 201 | 39 | 9 | 249
Age, Continuous [Median (Standard Deviation); unit: Months] | 32.03 (22.22) | 34.70 (22.12) | 13.26 (8.70) | 31.78 (22.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 23 | 5 | 147
  Male | 82 | 16 | 4 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 3 | 0 | 30
  Not Hispanic or Latino | 168 | 35 | 8 | 211
  Unknown or Not Reported | 6 | 1 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 31 | 5 | 1 | 37
  White | 142 | 29 | 7 | 178
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 25 | 3 | 1 | 29

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS)
Description: Probability of no relapse, secondary malignancy, or death whichever occurs first
Time Frame: 4 years from study enrollment
Population: All eligible BWT patients. 6 patients were excluded due to ineligibility and 6 patients were excluded due to protocol violation.
Measure: Mean (95% Confidence Interval); unit: Probability
Arm/Group | Arm 1 (Bilateral Wilms Tumors)
Number analyzed (Participants) | 189
Probability | 0.82 [0.74 to 0.91]

2. Primary Outcome: Kidney Preservation After Preoperative Chemotherapy
Description: Prevention of complete removal of at least one kidney in 50% of patients with bilateral Wilms tumor (BWT).
Time Frame: 12 weeks from study entry
Population: Eligible and evaluable Bilateral Wilms Tumor patients who completed pre-nephrectomy chemotherapy (VAD). 49 patients who did not complete VAD were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm 1 (Bilateral Wilms Tumors)
Number analyzed (Participants) | 140
Percentage of patients | 39 [31 to 47]

3. Primary Outcome: Number of Patients Without Complete Removal of at Least One Kidney
Description: To evaluate the efficacy of chemotherapy in preserving renal units in children with diffuse hyperplastic perilobar nephroblastomatosis (DHPLN) and preventing Wilms tumor development.
Time Frame: 12 weeks from the study entry
Population: Eligible and evaluable patients with diffuse hyperplastic perilobar nephroblastomatosis (DPHLN).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 3 (DHPLN)
Number analyzed (Participants) | 9
Participants | 7

4. Primary Outcome: Percentage of Patients Who Experienced Partial Nephrectomy After Preoperative Chemotherapy
Description: Percentage of patients who experienced partial nephrectomy in lieu of nephrectomy in 25% of children with unilateral tumors and aniridia, Beckwith-Wiedemann syndrome (BWS), hemihypertrophy or other overgrowth syndromes, by using prenephrectomy 2-drug chemotherapy induction with vincristine and dactinomycin.
Time Frame: 12 weeks from study entry
Population: Eligible and evaluable patients with unilateral high risk tumors who had partial or complete nephrectomy. 16 total patients were excluded (1 ineligible, 1 inevaluable, 1 violated protocol, and 13 did not have definitive surgery (partial or complete nephrectomy).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 2 (Unilateral High Risk Tumors Bilaterally Predisposed)
Number analyzed (Participants) | 23
percentage of patients | 57 [37 to 77]

5. Primary Outcome: Percentage of Patients Who Had Definitive Surgical Treatment
Description: Percentage of Bilateral Wilms Tumor (BWT) patients who undergo definitive surgery by week 12 after initiation of chemotherapy.
Time Frame: 12 weeks from study entry
Population: Eligible and evaluable Bilateral Wilms Tumor patients. 6 patients were excluded due to ineligible and 6 patients were excluded due to protocol violation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (Bilateral Wilms Tumors)
Number analyzed (Participants) | 189
percentage of participants | 85 [80 to 90]

ADVERSE EVENTS:
Time Frame: From enrollment to up to 10 years of follow-up
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Arm 1 (Bilateral Wilms Tumors) | Arm 2 (Unilateral High Risk Tumors Bilaterally Predisposed) | Arm 3 (DHPLN)
All-Cause Mortality (participants affected / at risk) | 10/189 | 0/36 | 0/9
Serious Adverse Events (participants affected / at risk) | 12/189 | 1/36 | 0/9
Other Adverse Events (participants affected / at risk) | 34/189 | 1/36 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Bilateral Wilms Tumors) (N=189) | Arm 2 (Unilateral High Risk Tumors Bilaterally Predisposed) (N=36) | Arm 3 (DHPLN) (N=9)
11600-Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
15000-Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
24600-Death NOS (General disorders) | 8 (8) | 0 (0) | 0 (0)
40600-Hepatobiliary disorders - Other specify (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0)
43100-Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
71500-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
83600-Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Bilateral Wilms Tumors) (N=189) | Arm 2 (Unilateral High Risk Tumors Bilaterally Predisposed) (N=36) | Arm 3 (DHPLN) (N=9)
10300-Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
10700-Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
11100-Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
11600-Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
11900-Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
13200-Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
14000-Aphonia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
14100-Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
15000-Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (2) | 0 (0)
15400-Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
18800-Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
20100-Cardiac disorders - Other specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
23400-Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
24100-Creatinine increased (Investigations) | 4 (6) | 0 (0) | 0 (0)
24700-Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
27800-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
28600-Ejection fraction decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
33300-Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0)
41400-Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
41600-Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
42100-Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
42500-Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
42700-Hypocalcemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
42900-Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
43100-Hypokalemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1) | 0 (0)
43200-Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
43500-Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
43900-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
50700-Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
51300-Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
58300-Neutrophil count decreased (Investigations) | 6 (8) | 0 (0) | 0 (0)
63900-Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
65800-Platelet count decreased (Investigations) | 2 (4) | 0 (0) | 0 (0)
66300-Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
68700-Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
71000-Renal and urinary disorders - Other specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
71500-Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
72500-Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
73700-Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
75700-Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
78100-Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
78900-Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
79600-Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
83100-Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
83600-Urine output decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
87900-Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
88500-White blood cell decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No